CLINICAL TRIAL: NCT06441331
Title: A Multicenter, Open-label, Interventional Phase I Trial to Determine the Dose and Evaluate the Pharmacokinetics (PK) and Safety of Lutetium Lu 177 Edotreotide Targeted Radiopharmaceutical Therapy (RPT) as Monotherapy or Following Standard of Care (SoC) for the Treatment of Somatostatin Receptor-positive Tumors in the Pediatric Population (KinLET).
Brief Title: Phase I Trial to Determine the Dose and Evaluate the PK and Safety of Lutetium Lu 177 Edotreotide Therapy in Pediatric Participants With SSTR-positive Tumors
Acronym: KinLET
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ITM Solucin GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITM-1191-01
Record Dates: First submitted 2024-05-22; First posted 2024-06-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Somatostatin Receptor Positive; NETs; Lymphoma; Solid Tumor; CNS Tumors; Rhabdomyosarcoma; Peripheral Primitive Neuroectodermal Tumor; GIST
Keywords: Pediatric; CNS tumors; Solid tumors; Lymphoma; Somatostatin Receptor (SSTR)-positive Tumors; Lutetium Lu 177 Edotreotide; Targeted RPT; ITM; GEP-NET; Neuroendocrine tumors; Radiopharmaceutical Therapy; Childhood
MeSH Terms: conditions — Lymphoma; Central Nervous System Neoplasms; Rhabdomyosarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Gastro-enteropancreatic neuroendocrine tumor; Neuroendocrine Tumors | interventions — 177Lu-octreotide, DOTA(0)-Tyr(3)-; amino-acid, glucose, and electrolyte solution

STUDY DESIGN:
Intervention Model Description: Three sequential age cohorts:
  1. ≥ 12 to < 18 years old
  2. ≥ 6 years to < 12 years old
  3. ≥ 2 to < 6 years old
  A minimum of 20 participants with SSTR-positive tumors of which at least six participants will have gastroenteropancreatic neuroendocrine tumors (GEP-NETs).
  A minimum of six participants will be required in each age cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Three sequential age cohorts (Experimental): Arms are based upon age at enrollment. The opening of the 2nd and 3rd cohort will depend on the recruitment of at least four participants with dosimetry and safety data for cycle 1, in the previous cohort.
  1. ≥ 12 to < 18 years old
  2. ≥ 6 years to < 12 years old
  3. ≥ 2 to < 6 years old
  Interventions: Drug: Lutetium Lu 177-Edotreotide; Other: Amino Acid Solution

INTERVENTIONS:
Drug: Lutetium Lu 177-Edotreotide — lutetium Lu 177 edotreotide At least two cycles and a maximum of six cycles at eight-week (± 2 we-ek) intervals. Extrapolation from standard maximum adult dose of 100 Megabecquerel(MBq)/kg for a 75 kg adult for the first cohort. Dosing decision for the subsequent cohorts by Data Monitoring Committee (DMC), based on (at least) cycle 1 dosimetry and safety data from at least four participants of the preceding cohort. Route of administration: Intravenous (IV) infusion. Duration of treatment: 16-48 weeks
  Other Names: 177Lu-edotreotide
Other: Amino Acid Solution — The Amino-Acid Solution (AAS) to be used in this study will contain a mixture of lysine and arginine diluted in an electrolyte solution.
  Other Names: Arginine-Lysine Solution

SUMMARY:
The purpose of the study is to determine the appropriate pediatric dosage and evaluate the pharmacokinetics (PK) and safety of Lutetium Lu 177 Edotreotide Targeted Radiopharmaceutical Therapy (RPT) as a monotherapy or following standard of care (SoC) in participants ≥2 to <18 years of age with somatostatin receptor (SSTR)-positive tumors.

DETAILED DESCRIPTION:
Determine the dose, pharmacokinetics and safety of Lutetium Lu 177 Edotreotide as monotherapy or following sequential standard of care in pediatric participants with recurrent, progressive or refractory NET, CNS, lymphoma and other solid tumors that express SSTRs by immunohistochemistry and demonstrate uptake by somatostatin receptor imaging. Lutetium Lu 177 Edotreotide will be given intravenously once every 8 weeks for a total of up to 6 doses over an average of 48 weeks in participants aged 2-18 years.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants aged ≥ 2 years and < 18 years
* Confirmed diagnosis somatostatin receptor-positive (SSTR-positive) disease.
* Tumor which is relapsed or is refractory to at least one line of previous therapy
* Positive SSTR protein expression confirmed by immunohistochemistry of a tumor histology sample
* Radioactivity uptake within the primary tumor or metastatic tumor sites measured by locally available SRIs ( 111In-based, 99mTc-based, or 68Ga-based SSTR single-photon emission computed tomography (SPECT)/ computed tomography (CT) or positron emission tomography (PET)/CT imaging, which is higher than the liver uptake)
* Participants must have recovered from the acute treatment related toxicities (defined as ≤ grade 1 if not defined in eligibility criteria, excluding alopecia, stable treated electrolyte abnormalities on replacement and stable treated hypothyroidism) of all prior treatment modality prior to entering this trial
* In case of sequential treatment followed by SoC or prior therapy, washout period applies before starting targeted RPT

Screening Consent Participant/legal guardian is willing to sign a screening consent. The screening consent is to be obtained according to institutional guidelines. Assent, when appropriate, will be obtained according to institutional guidelines.

Key Exclusion Criteria:

* Known hypersensitivity to Lutetium Lu 177 Edotreotide, DOTA/Edotreotide, or excipients
* Previous history of acute leukemia unless in remission for at least two years
* Extensive bone/bone marrow involvement as per Investigator's judgement unless peripheral blood stem cells (PBSC) are available at a minimum of 2.5x106 CD34+ cells/kg
* Patients who have received previous systemic targeted RPT
* Previous treatment with metaiodobenzyl guanidine (MIBG) if the predicted overall exposure is expected to exceed 2 Gy (gray) to the bone marrow or 23 Gy to the kidney.
* Previous treatment with external beam radiation therapy (EBRT) if the predicted overall exposure is expected to exceed more than 2 Gy to the bone marrow or 23 Gy to the kidney.
* Previous treatment with oncologic immune vaccine or CAR-T cell therapy
* Bulky disease in the CNS
* Presence of severe renal, hepatic, electrolyte, cardiovascular, or hematological dysfunction
* Participants who have received a live-attenuated vaccine up to four weeks prior to enrolment
* Pregnant or breastfeeding women.
* Other known malignancies.
* Serious non-malignant disease.

Ages: 24 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2034-04 (Estimated)

PRIMARY OUTCOMES:
Pediatric Dosage | a. Dosimetry assessments will be performed at multiple timepoints in cycle 1, 2 and 4. - b. Minimum of eight weeks after the first administration of Lutetium Lu 177 edotreotide
  Pediatric dosage based on:
  1. absorbed dose by target organs (kidney and bone marrow).
  2. rate of Dose limitting toxicities - based on adverse event reporting.

SECONDARY OUTCOMES:
Objective Response Rate | At the end of Cycle 2 (each cycle is 28 days)
  Assess preliminary anti-tumor activity by tumor type
PK and dosimetry | Dosimetry assessments will be performed at multiple timepoints at Cycle 1, 2 and 4.
  Lutetium Lu 177 edotreotide PK evaluation and tumor and target organ dosimetry
Rate of adverse events | From treatment start until 33 days following the last dose of trial treatment or until the End of Last Treatment (EOLT) visit, whichever occurs later..
  Safety evaluation of Lutetium Lu 177 edotreotide targeted RPT as monotherapy or following standard of care
Overall Survival, Progression-Free Survival and Duration of Response | Every 9 ± 3 weeks from enrollment until disease progression or for up to two years, whichever came first.
  Additional preliminary efficacy evaluation of lutetium Lu 177 Edotreotide targeted RPT as monotherapy or following SoC

OTHER OUTCOMES:
Exploratory Endpoint: Quality of Life | At enrollment, 18 days prior to cycles 2-6, four ± 3 weeks after targeted RPT.
  Assess quality of life based on the adapted Quality of Life (QoL) scale (PedsQL TM 3.0 Cancer Module)
Exploratory Endpoint: Correlation between SSTR expression detected by immunohisto-chemistry and functional imaging | No timeframe given.
  Correlation of the expression level of SSTR immunohistochemistry in tumor biopsy or surgery samples and 111In-based, 99mTc-based, or 68Ga-based-based lesion uptake (regarding intensity/distribution)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Henkel, PhD, Study Director — Director, Global Clinical Operations
Locations (2):
- The Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania, United States
- Hospital Universitario Vall d'Hebron - Oncología Médica, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No